CLINICAL TRIAL: NCT04921774
Title: Research on the Pathogenesis and Early Diagnosis of Acute Rejection in Patients With Heart Transplantation by Using Multimodality MR Imaging Combined With Circulating Exosomal miRNA Expression
Brief Title: Research on Patients With Heart Transplantation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Guangdong Provincial People's Hospital
Other Study IDs: 81771799
Record Dates: First submitted 2021-06-01; First posted 2021-06-10 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Heart Transplant Rejection
Keywords: Magnetic Resonance Imaging; Multimodality; Heart Transplantation; Exosome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This trial was a single-center, prospective cohort study.The purpose of this clinical research is to evaluate the accuracy of combining multimodality MR Imaging with circulating exosomal miRNA expression to diagnose acute rejection in patients with heart transplantation，thus it may be helpful for timely intervention to improve the patient's prognosis.

DETAILED DESCRIPTION:
Acute rejection (AR) after heart transplantation remains the major factor limiting long-term survival, and an independent risk factor for chronic allograft vasculopathy. Currently, there remains no reliable non-invasive method to detect AR. Multimodality magnetic resonance (MR) imaging shows accurate detection of myocardial damage, such as interstitial cell infiltrates, edema, hemorrhage, myocyte damage/necrosis and capillary stenosis or fragmentation. It turned out that the indicators in both MR imaging and circulating exosomal miRNA showed difference between patients with and without AR in our initial research work. Therefore, we hypothesize that circulating exosomal miRNA may play an important role in the activation of signaling pathway in AR after heart transplantation, which can be detected by multimodality MR imaging. All transplant recipients receiving transplantation follow-up care in our center were approached. In the present research we aim to combine multimodality MR imaging with circulating exosomal miRNA to explore a new evaluation methodology and platform for early and noninvasive detection of AR after heart transplantation. We attempt to confirm contribution of circulating exosomal miRNA to myocardial damage of AR through biopsy-proven allograft rejection and animal heterotopic heart transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. All patients after orthotopic heart transplantation.
2. All patients has signed informed consent.

Exclusion Criteria:

1. Patients with early graft failure within 24-48h after transplantation requiring clinical support or intensive care treatment.
2. Patients with severe renal failure.
3. Patients with any general contraindication to MRI.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients after orthotopic heart transplantation.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of combining multimodality MR Imaging with circulating exosomal miRNA expression in evaluating acute rejection in patients with heart transplantation. | At 6 months after surgery
  defined as the model's capability of accurately identifying patients who will have acute rejection.

SECONDARY OUTCOMES:
Specificity of combining multimodality MR Imaging with circulating exosomal miRNA expression in evaluating acute rejection in patients with heart transplantation. | At 6 months after surgery
  defined as the model's capability of accurately identifying patients who will not have acute rejection.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China